CLINICAL TRIAL: NCT04214288
Title: SERENA-2: A Randomised, Open-Label, Parallel-Group, Multicentre Phase 2 Study Comparing the Efficacy and Safety of Oral AZD9833 Versus Fulvestrant in Women With Advanced ER-Positive HER2-Negative Breast Cancer
Brief Title: A Study to Investigate Efficacy and Safety With Oral AZD9833 Compared With Intramuscular Fulvestrant in Post-menopausal Women at Least 18 Years of Age With Advanced ER-positive HER2 Negative Breast Cancer
Acronym: SERENA-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8530C00002; 2023-504974-40-00 (Registry Identifier: CTIS (EU)); 2019-003706-27 (EudraCT Number)
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced ER-Positive HER2-Negative Breast Cancer
Keywords: Open-Label; Parallel-Group; Fulvestrant; ER-Positive HER2-Negative Breast Cancer; Metastatic; AZD9833; Oral SERD; Camizestrant
MeSH Terms: conditions — Neoplasm Metastasis | interventions — AZD9833; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD9833 Dose A (Experimental): The patients will receive AZD9833 (Dose A).
  Interventions: Drug: AZD9833
- AZD9833 Dose B (Experimental): The patients will receive AZD9833 (Dose B).
  Interventions: Drug: AZD9833
- AZD9833 Dose C (Experimental): The patients will receive AZD9833 (Dose C).
  Interventions: Drug: AZD9833
- Fulvestrant 500 mg (Active Comparator): The patients will receive Fulvestrant (500 mg).
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD9833 — Dosage formulation: AZD9833 tablets will be administered orally.
  Arms: AZD9833 Dose A; AZD9833 Dose B; AZD9833 Dose C
Drug: Fulvestrant — Dosage formulation: Fulvestrant will be administered via intramuscular (IM) injection.
  Arms: Fulvestrant 500 mg

SUMMARY:
This study is randomized, open-label, parallel-group, multicentre Phase 2 study aimed to compare the efficacy and safety of oral AZD9833 versus intramuscular (IM) fulvestrant in women with advanced breast cancer.

DETAILED DESCRIPTION:
Post-menopausal women with histologically or cytologically confirmed metastatic or loco-regionally recurrent ER-positive HER2-negative breast cancer before randomization and fulfilling all of the inclusion criteria and none of the exclusion criteria will be included.

After the screening visit and confirmation of eligibility, patients will be randomly assigned in a 1:1:1:1 ratio to receive 1 of the following 4 treatments, consisting of 4-week treatment cycles until disease progression (assessed by the Investigator as defined by Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1):

* AZD9833 (Dose A)
* AZD9833 (Dose B)
* AZD9833 (Dose C)
* Fulvestrant (500 mg) During the treatment period, patients will have scheduled visits until treatment discontinuation. After the end of treatment, patients will attend 2 safety follow-up visits (at the time of treatment discontinuation and 28 days later) and will continue to be followed for survival.

As of December 2020, the Sponsor stopped enrolment to Dose C.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female patients aged at least 18 years.
* Metastatic or loco-regionally recurrent ER-positive HER2-negative adenocarcinoma of the breast.
* Radiological or other objective evidence of progression on or after the last systemic therapy prior to starting study treatment.
* Patients must have at least 1 lesion, not previously irradiated, that can be measured accurately at baseline as ≥10 mm in the longest diameter or in absence of measurable disease as defined above, at least 1 lytic or mixed (lytic+sclerotic) bone lesion.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organisation (WHO) performance status 0 to 1.
* Prior endocrine therapy as follows:

  1. Recurrence or progression on at least one line of endocrine therapy
  2. No more than 1 line of endocrine therapy for advanced disease
  3. No more than 1 line of chemotherapy for advanced disease
  4. Prior treatment with CDK4/6 inhibitors is permitted
  5. No prior treatment with fulvestrant, oral selective oestrogen receptor degrader (SERD), or related therapies
* Inclusion criterion for the paired tumour biopsy research subgroup:

Washout from prior tamoxifen: 4 months to elapse from last tamoxifen dose to pre-dose on-study biopsy.

Exclusion Criteria:

Intervention with any of the following:

* Any cytotoxic chemotherapy, investigational agents or other anti-cancer drugs for the treatment of breast cancer from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
* Use of systemic oestrogen-containing hormone replacement therapy within 6 months prior to the first dose of study treatment.
* Medications or herbal supplements known to be strong inhibitors/inducers of cytochrome P450 3A4/5 and sensitive CYP2B6 substrates, and drugs which are substrates of CYP2C9 and/or CYP2C19 which have a narrow therapeutic index or inability to stop use within the washout period prior to receiving the first dose of study treatment.
* Drugs that are known to prolong QT and have a known risk of torsades de pointes.
* The following cardiovascular criteria: QTcF >470 ms, resting heart rate <45 bpm, clinically significant abnormalities of resting electrocardiogram, uncontrolled hypertension, symptomatic hypotension, factors that increase the risk for QTc prolongation, left ventricular ejection fraction <50%.
* Radiotherapy with a limited field of radiation for palliation within 1 week of dosing, or to > 30% of bone marrow or a wide field within 4 weeks of dosing.
* Major surgical procedure or significant traumatic injury.
* Presence of life-threatening metastatic visceral disease or uncontrolled central nervous system metastatic disease.
* Inadequate bone marrow reserve or organ function.
* Refractory nausea and vomiting, uncontrolled chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9833.
* History of hypersensitivity to active or inactive excipients of AZD9833 or fulvestrant.
* Previous randomisation in the present study.
* Women of childbearing potential.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (9):
  - Research Site, Birmingham, Alabama
  - Research Site, Long Beach, California
  - Research Site, Fort Myers, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Lincoln, Nebraska
  - Research Site, Canton, Ohio
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Eagle River, Wisconsin
- Belgium (7):
  - Research Site, Brasschaat
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Haine-Saint-Paul
  - Research Site, Leuven
  - Research Site, Libramont-Chevigny
  - Research Site, Namur
- Canada (2):
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- France (2):
  - Research Site, Paris
  - Research Site, Vandœuvre-lès-Nancy
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (3):
  - Research Site, Berlin
  - Research Site, Düsseldorf
  - Research Site, Essen
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
- Italy (9):
  - Research Site, Bologna
  - Research Site, Catanzaro
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Umbria
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Piła
  - Research Site, Rzeszów
  - Research Site, Skorzewo
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Almada
  - Research Site, Lisbon
- Russia (8):
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Incheon
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Zaragoza
- Ukraine (6):
  - Research Site, Cherkasy
  - Research Site, Chernivtsі
  - Research Site, Kyiv
  - Research Site, M. Kyiv
  - Research Site, S. Khodosivka
  - Research Site, Uzhhorod
- United Kingdom (2):
  - Research Site, Derby
  - Research Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Oliveira M, Pominchuk D, Nowecki Z, Hamilton E, Kulyaba Y, Andabekov T, Hotko Y, Melkadze T, Nemsadze G, Neven P, Vladimirov V, Zamagni C, Denys H, Forget F, Horvath Z, Nesterova A, Ajimi M, Kirova B, Klinowska T, Lindemann JPO, Lissa D, Mathewson A, Morrow CJ, Traugottova Z, van Zyl R, Arkania E. Camizestrant, a next-generation oral SERD, versus fulvestrant in post-menopausal women with oestrogen receptor-positive, HER2-negative advanced breast cancer (SERENA-2): a multi-dose, open-label, randomised, phase 2 trial. Lancet Oncol. 2024 Nov;25(11):1424-1439. doi: 10.1016/S1470-2045(24)00387-5. PMID 39481395
- [Derived] Hamilton E, Oliveira M, Turner N, Garcia-Corbacho J, Hernando C, Ciruelos EM, Kabos P, Ruiz-Borrego M, Armstrong A, Patel MR, Vaklavas C, Twelves C, Boni V, Incorvati J, Brier T, Gibbons L, Klinowska T, Lindemann JPO, Morrow CJ, Sykes A, Baird RD. A phase I dose escalation and expansion trial of the next-generation oral SERD camizestrant in women with ER-positive, HER2-negative advanced breast cancer: SERENA-1 monotherapy results. Ann Oncol. 2024 Aug;35(8):707-717. doi: 10.1016/j.annonc.2024.04.012. Epub 2024 May 8. PMID 38729567
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00002&attachmentIdentifier=8b692168-dc6e-4f1d-8150-3681e326e2e3&fileName=D8530C00002_CSP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00002&attachmentIdentifier=1fab540e-32f7-4db8-823d-75b90ee044f7&fileName=D8530C00002_SAP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8530C00002&attachmentIdentifier=d319ed5c-8795-4684-8602-d1e34032181f&fileName=D8530C00002_CSRSynopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were enrolled at 82 sites in 16 countries from 22 April 2020 to 30 August 2022. The study is ongoing.
Groups:
- AZD9833 75mg: The patients received AZD9833 75mg oral tablets once daily.
- AZD9833 150mg: The patients received AZD9833 150mg oral tablets once daily.
- AZD9833 300mg: The patients received AZD9833 300mg oral tablets once daily.
- Fulvestrant 500 mg: The patients received Fulvestrant 500 mg via Intramuscular (IM) injection.
Period: Overall Study
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
Started | 74 | 73 | 20 | 73
Completed | 0 | 0 | 0 | 0
Not Completed | 74 | 73 | 20 | 73
Not completed — Ongoing in the study | 41 | 51 | 12 | 39
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 22 | 13 | 7 | 19
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0
Not completed — Other | 1 | 2 | 0 | 6
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 0 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all randomised patients, with treatment groups assigned in accordance with the randomisation, regardless of the actual treatment received.
Groups:
- Fulvestrant 500 mg: The patients received Fulvestrant 500 mg via IM injection.
- Total: Total of all reporting groups
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg | Total
Number analyzed (Participants) | 74 | 73 | 20 | 73 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (9.56) | 61.7 (9.68) | 59.9 (10.72) | 59.3 (11.08) | 60.7 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 73 | 20 | 73 | 240
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 71 | 70 | 20 | 65 | 226
  Other | 3 | 3 | 0 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was assessed by the Investigator as defined by response evaluation criteria in solid tumors (RECIST) version 1.1. PFS was defined as the time from randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from randomised therapy or received another anti-cancer therapy prior to progression. Disease progression was defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
  Data from the 300mg arm should be interpreted with caution as recruitment to the 300mg arm was stopped early at 20 patients randomised and therefore the 300mg data is highly variable.
Time Frame: From date of randomisation to date of objective disease progression (or last evaluable assessment in the absence of progression) or death (up to data cut-off of 29 months)
Population: FAS consisted of all randomised patients, with treatment groups assigned in accordance with the randomisation, regardless of the actual treatment received.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
Number analyzed (Participants) | 74 | 73 | 20 | 73
Months | 7.2 [3.7 to 10.9] | 7.7 [5.5 to 12.9] | 6.3 [1.9 to NA] — The upper limit of 90% confidence interval (CI) was not estimable due to insufficient data. | 3.7 [2.0 to 6.0]
Statistical Analysis 1: Comparison: AZD9833 75mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.0167, Log Rank; The analysis was performed using a stratified Cox Proportional Hazards model; Hazard Ratio (HR) = 0.59, 90% CI [0.42 to 0.82] — A hazard ratio < 1 favours AZD9833 to be associated with a longer progression-free survival than fulvestrant
Statistical Analysis 2: Comparison: AZD9833 150mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.0090, Log Rank; The analysis was performed using a stratified Cox Proportional Hazards model; Hazard Ratio (HR) = 0.64, 90% CI [0.46 to 0.89] — A hazard ratio < 1 favours AZD9833 to be associated with a longer progression-free survival than fulvestrant

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was assessed by the Investigator as defined by RECIST version 1.1. The ORR was defined as investigator assessed Complete Response or Partial Response prior to progression in patients with measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
  Adjusted response rate was presented in this analysis.
  Data from the 300mg arm should be interpreted with caution as recruitment to the 300mg arm was stopped early at 20 patients randomised and therefore the 300mg data is highly variable.
Time Frame: From screening until disease progression (up to data cut-off of 29 months)
Population: A subset of the FAS with measurable disease.
Measure: Number; unit: Percentage (%)
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
Number analyzed (Participants) | 70 | 65 | 19 | 68
Percentage (%) | 15.7 | 17.1 | 25.2 | 11.6
Statistical Analysis 1: Comparison: AZD9833 75mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.4828, Regression, Logistic; The analysis was performed using logistic regression model adjusting for prior use of CDK4/6 inhibitors and presence of lung and/or liver metastasis; Odds Ratio (OR) = 1.42, 90% CI [0.63 to 3.31] — An odds ratio > 1 favours AZD9833
Statistical Analysis 2: Comparison: AZD9833 150mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.3691, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.57, 90% CI [0.69 to 3.67] — An odds ratio > 1 favours AZD9833

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR was assessed by the Investigator as defined by RECIST version 1.1. The DoR was defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression.
Time Frame: From screening until disease progression or last evaluable assessment in the absence of progression (up to data cut-off of 29 months)
Reporting Status: Not Posted, anticipated posting 2027-03

4. Secondary Outcome: Percentage Change in Tumour Size at 16 Weeks
Description: The percentage change in tumour size at 16 weeks was obtained for each patient, based on RECIST measurements taken at baseline and at 16 weeks. Tumour size is the sum of the longest diameters of the target lesions (TLs). Percentage change in the sum of longest TLs diameters at 16 weeks was measured.
Time Frame: At Week 16
Reporting Status: Not Posted, anticipated posting 2027-03

5. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from randomisation to death due to any cause.
Time Frame: From the date of randomisation until death (up to data cut-off of 29 months)
Reporting Status: Not Posted, anticipated posting 2027-03

6. Secondary Outcome: Clinical Benefit Rate at 24 Weeks (CBR24)
Description: Clinical benefit rate was defined as patients with best objective response of complete response or partial response in the first 25 weeks or who have stable disease for at least 23 weeks after randomization.
  Adjusted response rate was presented in this analysis.
  Data from the 300mg arm should be interpreted with caution as recruitment to the 300mg arm was stopped early at 20 patients randomised and therefore the 300mg data is highly variable.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage (%)
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
Number analyzed (Participants) | 74 | 73 | 20 | 73
Percentage (%) | 48.8 | 51.0 | 42.4 | 39.1
Statistical Analysis 1: Comparison: AZD9833 75mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.2554, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.48, 90% CI 2-sided [0.84 to 2.64] — An odds ratio > 1 favours AZD9833
Statistical Analysis 2: Comparison: AZD9833 150mg vs Fulvestrant 500 mg; Test type: Superiority; p = 0.1658, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.62, 90% CI [0.91 to 2.89] — An odds ratio > 1 favours AZD9833

7. Secondary Outcome: Plasma Concentrations of AZD9833
Description: The plasma concentrations of AZD9833 at steady state were evaluated.
Time Frame: Cycle 1 Day 15 (pre-dose), Cycle 1 Day 15 (2h), Cycle 1 Day 15 (4h) and Cycle 2 Day 1 (pre-dose), (each cycle is 28 days in length)
Population: The PK Analysis Set consisted of all patients who received at least one dose of AZD9833 per protocol, for whom there is at least one reportable PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg
Number analyzed (Participants) | 69 | 68 | 19
ng/ml
  Cycle 1 Day 15 (pre-dose): number analyzed (Participants) | 69 | 67 | 18
  Cycle 1 Day 15 (pre-dose) | 22.8387 (84.3207) | 41.0856 (148.5806) | 108.1351 (157.3080)
  Cycle 1 Day 15 (2h): number analyzed (Participants) | 69 | 64 | 18
  Cycle 1 Day 15 (2h) | 51.9098 (94.4632) | 96.2038 (164.5328) | 302.1254 (66.9155)
  Cycle 1 Day 15 (4h): number analyzed (Participants) | 69 | 62 | 19
  Cycle 1 Day 15 (4h) | 54.5098 (87.2152) | 95.5360 (160.0032) | 289.1464 (68.1607)
  Cycle 2 Day 1 (pre-dose): number analyzed (Participants) | 64 | 68 | 18
  Cycle 2 Day 1 (pre-dose) | 24.2895 (88.4140) | 34.2592 (245.9897) | 115.8558 (156.4858)

8. Secondary Outcome: Percent Change From Baseline in ER and PgR Expression and Ki67 Labelling Index
Description: The pharmacodynamics of AZD9833 and fulvestrant in a subgroup of patients.
Time Frame: From baseline to Cycle 2 Day 1 (each cycle is 28 days in length)
Reporting Status: Not Posted, anticipated posting 2027-03

9. Secondary Outcome: Changes From Baseline in Health Related Quality of Life (HRQoL)
Description: To evaluate the effect of AZD9833 and fulvestrant on the patients' health-related quality of life, as assessed by patient completed HRQoL questionnaires.
Time Frame: From Day 1 until end of treatment and safety follow up (up to data cut-off of 29 months)
Reporting Status: Not Posted, anticipated posting 2027-03

10. Other Pre Specified Outcome: Number of Patients With Adverse Events
Description: The safety and tolerability of AZD9833 when compared to fulvestrant in women with advanced ER-positive HER2-negative breast cancer was evaluated.
Time Frame: From the date of first dose up to the safety follow-up period (28 days after last dose of AZD9833 and 56 days after last dose of fulvestrant) (up to data cut-off of 29 months)
Population: Safety analysis set consisted of all patients who received any amount of study treatment (AZD9833 or fulvestrant), regardless of whether that was the randomised therapy intended or whether they received therapy without being randomised and for whom any post-dose data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
Number analyzed (Participants) | 74 | 73 | 20 | 73
Participants
  Any Adverse Event (AE) | 57 | 66 | 19 | 50
  Any AE causally related to treatment | 39 | 49 | 14 | 13
  Any AE of CTCAE grade 3 or higher | 9 | 17 | 3 | 11
  Any AE of CTCAE grade 3 or higher, causally related to treatment | 1 | 2 | 1 | 0
  Any AE with outcome = death | 0 | 1 | 0 | 0
  Any AE with outcome = death, causally related to treatment | 0 | 0 | 0 | 0
  Any Serious Adverse Event (SAE) | 6 | 7 | 2 | 4
  Any SAE, causally related to treatment | 3 | 2 | 1 | 0
  Any SAE causing discontinuation of treatment | 1 | 0 | 0 | 0
  Any SAE causing discontinuation of treatment, causally related to treatment | 1 | 0 | 0 | 0
  Any AE leading to discontinuation of treatment | 2 | 0 | 2 | 0
  Any AE leading to discontinuation of treatment, causally related to treatment | 2 | 0 | 0 | 0
  Any AE leading to dose reduction | 1 | 9 | 4 | 0
  Any AE leading to dose interruption | 11 | 16 | 4 | 3

ADVERSE EVENTS:
Time Frame: From the date of first dose up to the safety follow-up period (28 days after last dose of AZD9833 and 56 days after last dose of fulvestrant) (up to data cut-off of 29 months)
Arm/Group | AZD9833 75mg | AZD9833 150mg | AZD9833 300mg | Fulvestrant 500 mg
All-Cause Mortality (participants affected / at risk) | 23/74 | 14/73 | 7/20 | 21/73
Serious Adverse Events (participants affected / at risk) | 6/74 | 7/73 | 2/20 | 4/73
Other Adverse Events (participants affected / at risk) | 44/74 | 61/73 | 17/20 | 31/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AZD9833 75mg (N=74) | AZD9833 150mg (N=73) | AZD9833 300mg (N=20) | Fulvestrant 500 mg (N=73)
Breast cellulitis (Infections and infestations) | 0 (0) | 1/7 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0/7 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1/7 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AZD9833 75mg (N=74) | AZD9833 150mg (N=73) | AZD9833 300mg (N=20) | Fulvestrant 500 mg (N=73)
COVID-19 (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (6) | 3 (4) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 11 (16) | 1 (1) | 5 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (5) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 3 (3) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 5 (6) | 6/72 (8) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Photopsia (Eye disorders) | 9 (11) | 18 (28) | 7 (10) | 0 (0)
Visual impairment (Eye disorders) | 5 (5) | 5 (5) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 12 (12) | 6 (8) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 4 (4) | 7 (10) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 6 (7) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 4 (4) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 9 (11) | 2 (2) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (3) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (4)
Asthenia (General disorders) | 6 (6) | 11 (13) | 2 (3) | 5 (5)
Fatigue (General disorders) | 4 (4) | 14 (19) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 2 (3) | 4 (4) | 0 (0) | 1 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 6 (10) | 3 (4) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 6 (10) | 2 (2) | 5 (6)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (3) | 1 (1) | 2 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
At the time of CSR finalization, CSP version 5.0 was available, therefore, CSP version 5.0 was redacted and submitted along with the Results Registration Form.

Data from the 300mg arm should be interpreted with caution as recruitment to the 300mg arm was stopped early at 20 patients randomised and therefore the 300mg data is highly variable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT04214288/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04214288/SAP_001.pdf